CLINICAL TRIAL: NCT04781426
Title: Pre-exposure Prophylaxis of HIV Infection Among Men Who Have Sex With Men (MSM) and Transgender Women (TG) in Suburban Yangon, Myanmar
Brief Title: PrEP Among MSM and TG in Myanmar
Acronym: PrEP
Status: Completed | Type: Observational
Sponsor: Myanmar Oxford Clinical Research Unit (Other)
Collaborators: Medical Action Myanmar (Other); Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: OXTREC 49-20
Record Dates: First submitted 2021-02-25; First posted 2021-03-04 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: HIV Infections
Keywords: Pre-exposure prophylaxis of HIV infection; PrEP; MSM; TG
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; Lamivudine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV-negative MSM/TG: Oral pre-exposure prophylaxis (PrEP) will be offered to HIV negative MSM, TG identified to be at substantial risk for HIV infection and those motivated to take daily PrEP.
  Interventions: Drug: Tenofovir Disoproxil Fumarate (TDF) 300 mg

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate (TDF) 300 mg — PrEP regimens of Tenofovir Disoproxil Fumarate (TDF) 300 mg/Lamivudine (3TC) 300mg per oral (PO) daily
  Other Names: Lamivudine (3TC) 300mg

SUMMARY:
HIV is concentrated among key populations in Myanmar. Globally, HIV-prevalence among transgender (TG) women is one of the highest; laboratory-confirmed prevalence is reported up to 40%. In September 2015, WHO recommended the use of Pre-Exposure Prophylaxis (PrEP) for people at substantial risk of HIV as part of a combination HIV prevention strategy. A demonstration project will take place to implement and evaluate the uptake and effectiveness of PrEP among MSM, and TG women in a clinic in Hlaingtharyar township, Yangon. The aim is to describe PrEP uptake, as well as HIV-seroconversion and STI infection rates among those who use PrEP.

ELIGIBILITY:
Inclusion Criteria:

* HIV-negative
* No suspicion of acute HIV infection
* Substantial risk of HIV infection
* Creatinine clearance is more than 30 ml/min
* Willingness to use PrEP as prescribed, including periodic HIV testing
* Willingness to sign informed consent

Exclusion Criteria:

• Anyone who is not eligible with the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals self-identified as belonging to the MSM and/or TG population who are eligible in line with selection criteria
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Uptake rate of PrEP | through study completion, an average of 1 year
  The proportion of HIV-negative MSM and TG women who are taking PrEP among those who are eligible to take PrEP.
HIV seroconversion rate among PrEP user | through study completion, an average of 1 year
  The portion of PrEP taking HIV negative MSM and TG women who become HIV positive while he is taking PrEP among those who are taking PrEP.
STI infection rates among PrEP user(Syphilis test, Gram stain for gonorrhoea and Xpert CT/NG) | through study completion, an average of 1 year
  The number of positive episodes for either syphilis or gonorrhea or chlamydia infection among the PrEP taking MSM and Transgender women per number of testing among them.

CONTACTS AND LOCATIONS:
Overall Officials: NiNi Tun, MB BS, Principal Investigator — Medical Action Myanmar
Locations (1):
- Medical Action Myanmar Clinics, Yangon, Burma

IPD SHARING:
Plan to Share IPD: Undecided